CLINICAL TRIAL: NCT04053140
Title: Closed-loop Control of Penicillin Delivery Integrating Electrochemical Biosensor Technology
Brief Title: Closed-loop Control of Penicillin Delivery
Acronym: CLCPD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 251161
Record Dates: First submitted 2019-07-24; First posted 2019-08-12 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Healthy Volunteers
Keywords: Pharmacokinetics; Penicillin G; Penicillins; Proof of Concept Study; Clinical Trial, Phase I; Microneedle array
MeSH Terms: interventions — Penicillin G

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Routine intermittent slow bolus (Experimental): The microneedle biosensor will be sited peripherally (on the non-dominant arm) for the duration of the study. It will then be removed. Benzylpenicillin IV 1200mg administered every 4 hours.
  Interventions: Device: Microneedle array; Drug: Penicillin G_1200mg
- Closed-loop control of intermittent slow bolus (Experimental): The microneedle biosensor will be sited peripherally (on the non-dominant arm) for the duration of the study. It will then be removed. Benzylpenicillin IV administered in intermittent dosing schedule. Dosage to be determined by closed-loop algorithm. Limits set to 2400mg every 4 hours.
  Interventions: Device: Microneedle array and closed-loop control of penicillin delivery; Drug: Penicillin G_2400mg
- Closed-loop control of continuous infusion (Experimental): The microneedle biosensor will be sited peripherally (on the non-dominant arm) for the duration of the study. It will then be removed. Benzylpenicillin IV administered in continuous dosing schedule. Dosage to be determined by closed-loop algorithm. Initial loading dose, and limits set to 600mg/hr.
  Interventions: Device: Microneedle array and closed-loop control of penicillin delivery; Drug: Penicillin G_600mg/hr

INTERVENTIONS:
Device: Microneedle array — The microneedle biosensor will be sited peripherally (on the non-dominant arm) for the duration of the study. It will then be removed.
  Arms: Routine intermittent slow bolus
Device: Microneedle array and closed-loop control of penicillin delivery — The microneedle biosensor will be sited peripherally (on the non-dominant arm) for the duration of the study. It will then be removed. Microneedle data will be used to titrate benzylpenicillin dosage according to PK-PD target.
  Arms: Closed-loop control of continuous infusion; Closed-loop control of intermittent slow bolus
Drug: Penicillin G_1200mg — Benzylpenicillin IV 1200mg administered every 4 hours.
  Other Names: Benzylpenicillin
  Arms: Routine intermittent slow bolus
Drug: Penicillin G_2400mg — Benzylpenicillin IV administered in intermittent dosing schedule. Dosage to be determined by closed-loop algorithm. Limits set to 2400mg every 4 hours.
  Other Names: Benzylpenicillin
  Arms: Closed-loop control of intermittent slow bolus
Drug: Penicillin G_600mg/hr — Benzylpenicillin IV administered in continuous dosing schedule. Dosage to be determined by closed-loop algorithm. Initial loading dose, and limits set to 600mg/hr.
  Other Names: Benzylpenicillin
  Arms: Closed-loop control of continuous infusion

SUMMARY:
This study is an in-house feasibility study of penicillin biosensor technology linked with closed-loop control for the automated delivery of penicillin antibiotics.

DETAILED DESCRIPTION:
Outline of the study:

This study will take place at the Imperial Clinical Research Facility (ICRF). Twenty healthy volunteers will be recruited to take part in three visits to the ICRF. These will each last 8-12 hours. During these visits participants will receive penicillin via infusion following:

(i) Routine (intermittent or continuous) dosing protocols. (ii) Intermittent dosing directed by a closed-loop control system. (iii) Continuous dosing directed by a closed-loop control system. Participants will have up to 15 blood samples and tissue microdialysis performed. A biosensor will also be used to provide real-time antibiotic concentration data. This will be used to drive the closed-loop control system. Outcome measures will be PK-PD target attainment between visits. This target will be 50% time > MIC and 100% time > MIC.

Participant identification:

Healthy volunteers will be recruited from a healthy volunteer database held within Imperial College London and via identification of participants within the College. An initial advertisement e-mail will be sent by the Healthy Volunteer Database Administrator and individuals responding will then followed up by telephone or e-mail and invited to attend a screening visit at the ICRF. They will be sent the participant information leaflet via email in advance of this meeting to give them time to consider the information.

Study methodology:

* Twenty healthy volunteers will be invited to participate in an exploratory study of the biosensor device and closed-loop control systems.
* Allergy status will be confirmed with the participant at each visit.
* Study days will follow the same format. The only deviation will be the method of penicillin delivery (this will either be by routine infusion, closed-loop intermittent infusion, or closed-loop continuous infusion).
* On the night before study visits, participants will be asked to refrain from drinking alcohol. On the study day they will be invited to bring a laptop / tablet device for their entertainment. Alternatively, one will be provided on the study day by the ICRF.
* On arrival at the study center the participant will have a microneedle biosensor sited.
* They will have two cannulae inserted, ideally one in each arm. One of these will be for taking blood during the study. The other will be for penicillin delivery.
* They will also have a microdialysis fibre inserted in the same arm as the microneedle array.
* A baseline blood sample will be taken (full blood count, renal function, liver function, and C-reactive protein) on each visit.
* The microneedle biosensor will be sited peripherally (on the non-dominant arm). These sensors are connected to potentiostat devices that record data, which can then be downloaded onto a computer for analysis.
* The study will then commence at time = 0 when the first infusion of penicillin will be given.
* In total, the study will run for 3 benzylpenicillin dosing intervals (8-12 hours). For intermittent, routine care benzylpenicillin doses will be given at time = 0, 4, and 8 hours. During closed-loop control visits the controller will be allowed to determine the dosing interval / period. The controller will be limited to deliver a MAXIMUM dose equivalent to 2.4g every 4-hours.
* During the study interval the participant will undergo rich blood and microdialysis drug concentration sampling. For blood sampling, up to 15 beta-lactam drug levels will be taken during the study visit period. Each blood test will involve the collection of 5mLs of blood (1 teaspoon). Microdialysis will be performed continuously for the study period. The collection vial will be changed every 15-30 minutes during the study period.
* In addition, a blood spot will be used from the blood samples taken as part of the PK sampling to test point-of-care penicillin sensors at the time-points described below.
* A visual analogue scale will be completed by the participant every hour to evaluate their level of discomfort due to the microneedle sensor device. The device and site will also be checked by researchers every hour.
* Time points for the blood sampling are planned to initially be taken at pre, 6, 10, 15, 30, 60, 120, 180, 240, 246, 250, 300, 480, 486, 600 minutes. However, following initial PK analysis a D-optimal design will be employed using Pmetrics and BestDose pharmacokinetic software to determine the optimal time points for blood PK analysis.

ELIGIBILITY:
Inclusion Criteria:

* Adult >18 years old.
* Healthy adults, with no evidence of infection.
* Previously received penicillin with no adverse effects.

Exclusion Criteria:

* < 18 years old.
* High risk of skin and soft tissue infection or local skin and soft tissue infection near sensor site.
* Hypersensitivity to adhesive strips or active dermatitis.
* Penicillin hypersensitivity or previous adverse event whilst receiving penicillin.
* Anaemia on screening bloods (defined as haemoglobin <13 g/dL in males and <12 g/dL in females).
* Renal impairment on screening bloods (defined as a Cockcroft-Gault creatinine clearance <60mL/min).
* Liver impairment on screening bloods (defined as ALT, ALP or bilirubin 3x ULN).
* Implantable electronic device in-situ if wearing a microneedle array device.
* Pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Assessment of the biosensors ability to track benzylpenicillin concentrations compared to observations made by microdialysis and blood sampling. | Up to 12 hours.
  Bland-Altman plot to describe agreement between interstitial benzylpenicillin concentrations and microneedle data.
Compare PK-PD target attainment between visits | Up to 12 hours.
  Compare time > MIC between visits

CONTACTS AND LOCATIONS:
Overall Officials: Alison H Holmes, MD MPH MBBS, Principal Investigator — Health Protection Research Unit in HCAI & AMR
Locations (1):
- NIHR Imperial CRF, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gowers SAN, Freeman DME, Rawson TM, Rogers ML, Wilson RC, Holmes AH, Cass AE, O'Hare D. Development of a Minimally Invasive Microneedle-Based Sensor for Continuous Monitoring of beta-Lactam Antibiotic Concentrations in Vivo. ACS Sens. 2019 Apr 26;4(4):1072-1080. doi: 10.1021/acssensors.9b00288. Epub 2019 Apr 17. PMID 30950598
- See also: Minimally Invasive Sensing of Beta-lactam Antibiotics (MISBL) — https://clinicaltrials.gov/ct2/show/NCT03847610